CLINICAL TRIAL: NCT02421848
Title: Body Composition Evaluation of Cirrhotic Patients With Ascites
Brief Title: Lean Mass Evaluation of Cirrhotic Patients With Ascites With the Use DXA
Acronym: BCECPA
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Dan Linetzky Waitzberg, Dan Linetzky Waitzberg, University of Sao Paulo
Other Study IDs: U São Paulo
Record Dates: First submitted 2015-03-26; First posted 2015-04-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Liver Cirrhosis
Keywords: Body composition; Sarcopenia; Cirrhotic with Ascites
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cirrhotic Patients With Ascites: Cirrhotic Patients With Ascites

SUMMARY:
Malnutrition due to liver disease is common, however, their detection is difficult. The parameters used for nutritional assessment in clinical practice have limited use in this patient population.

From this perspective, this study proposes to develop predictive equations for body composition for electrical bioimpedance (BIA) in cirrhotic patients. Besides being a fast and risk free, the BIA offers the additional advantage of low cost compared to other methods that assess body composition (BC).

Will be selected patients male with liver cirrhosis (n = 112) of the Liver Transplant Clinic of the Hospital of the Clinicas, Faculty of Medicine, University of São Paulo.

This pioneering study is of great clinical importance because malnutrition is a relevant factor in the prognosis of liver disease and there is not efficient method in clinical practice to properly assess the body composition in this population.

DETAILED DESCRIPTION:
Malnutrition due to liver disease is common, however, their detection is difficult. The parameters used for nutritional assessment in clinical practice have limited use in this patient population.

From this perspective, this study proposes to develop predictive equations for body composition for electrical bioimpedance (BIA) in cirrhotic patients. Besides being a fast and risk free, the BIA offers the additional advantage of low cost compared to other methods that assess body composition (BC).

Will be selected patients male with liver cirrhosis (n = 112) of the Liver Transplant Clinic of the Hospital of the Clinicas, Faculty of Medicine, University of São Paulo. After signing an informed consent, BC will be estimated by bioelectrical impedance analysis and by reference method (DXA). The data obtained by both methods are statistically treated to obtain specific BIA prediction equations for the evaluation of cirrhotic patients.

This pioneering study is of great clinical importance because malnutrition is a relevant factor in the prognosis of liver disease and there is not efficient method in clinical practice to properly assess the body composition in this population. Such knowledge, in turn, can serve as a new tool for nutritional assistance in treating this disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-60 years) of both sexes;
* Signing the free and informed consent;
* Show interest, conditions and availability to participate in all procedures included in the study protocol;
* liver cirrhosis Carrier

Exclusion Criteria:

* Refusal to participate;
* Patients who have made liver transplantation;
* Physical Amputation;
* Swelling in the lower limb;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will be selected patients male with liver cirrhosis (n = 112) of the Liver Transplant Clinic of the Hospital of the Clinicas, Faculty of Medicine, University of São Paulo.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body Composition Evaluation of Cirrhotic Patients With Ascites (estimated by bioelectrical impedance analysis and by reference method (DXA) | two years

REFERENCES:
- [Derived] Belarmino G, Singer P, Gonzalez MC, Machado NM, Cardinelli CS, Barcelos S, Andraus W, D'Albuquerque LAC, Damiani L, Costa AC, Pereira RMR, Heymsfield SB, Sala P, Torrinhas RSM, Waitzberg DL. Prognostic value of energy expenditure and respiratory quotient measuring in patients with liver cirrhosis. Clin Nutr. 2019 Aug;38(4):1899-1904. doi: 10.1016/j.clnu.2018.07.001. Epub 2018 Jul 6. PMID 30007480